CLINICAL TRIAL: NCT02536755
Title: Open Label Interventional Multicenter Phase 3b Study to Evaluate Skeletal Response to Eliglustat in Adult Patients Who Successfully Completed the Phase 2 or Phase 3 Studies
Brief Title: Phase 3b Study to Evaluate Skeletal Response to Eliglustat in Adult Patients Who Completed Phase 2 or Phase 3 Studies
Acronym: EXOSKEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC13781; U1111-1166-6190 (Other: UTN)
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eliglustat (Experimental): Participants who completed one of the Phase 2 (GZGD00304 [NCT00358150]) or Phase 3 studies (GZGD02507 [NCT00891202], GZGD02607 [NCT00943111], or GZGD03109 [NCT01074944]) were enrolled in this current (EFC13781) study. Participants who were cytochrome P450 (CYP) 2D6 intermediate metabolizer (IM), extensive metabolizer (EM) and ultra-rapid metabolizers (URM) received eliglustat 84 milligrams (mg) twice daily and participants who were CYP2D6 poor metabolizer (PM) received eliglustat 84 mg once daily, for duration of minimum 2 years (unless early discontinuation occurred) and up to 4 years, or until commercial eliglustat was available to participants through reimbursement or through the compassionate use (expanded access) program.
  Interventions: Drug: Eliglustat, GZ385660

INTERVENTIONS:
Drug: Eliglustat, GZ385660 — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: Cerdelga

SUMMARY:
Primary Objective:

Evaluate long term skeletal response to eliglustat in adult participants who successfully completed one of the Phase 2 or Phase 3 eliglustat studies.

Secondary Objective:

Evaluate the safety of eliglustat (by serious adverse event continuous monitoring), the quality of life (Short Form-36 Health Survey [SF-36]) and biomarkers of Gaucher disease type 1 (GD1) (chitotriosidase, plasma glucosylceramide [GL-1] and lyso glucosylceramide [lyso-GL-1]) in adult participants who successfully completed one of the Phase 2 or Phase 3 studies.

DETAILED DESCRIPTION:
Study duration for individual participants was to be of minimum 2 years and up to 4 years, or until commercial eliglustat was available to participants through reimbursement. If after 4 years since the beginning of the study eliglustat was not approved and available to participants in participating country, participants in this country might continue to receive study treatment until eliglustat was available to participants through the compassionate use (expanded access) program or was approved and available through reimbursement, whichever came first.

ELIGIBILITY:
Inclusion criteria :

* The participant must have successfully completed the Phase 2 (GZGD00304) or a Phase 3 study (GZGD02507, GZGD02607 or GZGD03109). Successful completion was defined as participants enrolled in one of the above mentioned studies who received eliglustat through the end of the study and completed the end-of-study visit without having discontinued or been withdrawn prematurely.
* The participant was willing and able to provide signed informed consent prior to any protocol-required procedures being performed.
* Female participants of childbearing potential must have had a documented negative pregnancy test prior to enrollment and while they were receiving eliglustat treatment.
* Female participants of childbearing potential must have been willing to practice true abstinence in line with their preferred and usual lifestyle, or used a medically accepted form of contraception (either a barrier method, such as condom or diaphragm + spermicide, or a non-barrier method such as oral, injected, or implanted hormonal methods, or an intra-uterine device or system) while receiving eliglustat.

Exclusion criteria:

* The participant was unwilling to comply with the requirements of the protocol.
* The participant had received an investigational product (other than eliglustat) within 30 days prior to enrollment.
* The participant had received miglustat within the 6 months prior to enrollment.
* The participant had documented prior esophageal varices or liver infarction or current liver enzymes (alanine transaminase, aspartate aminotransferase) or total bilirubin greater than (>)2 times the upper limit of normal, unless the participant had a diagnosis of Gilbert Syndrome.
* The participant had any clinically significant disease, other than Gaucher disease, including cardiovascular, renal, hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic (eg, hypokalemia, hypomagnesemia), or psychiatric disease, other medical conditions, or serious intercurrent illnesses that might preclude participation in the study.
* The participant was known to have any of the following: cardiac disease (congestive heart failure, recent acute myocardial infarction, bradycardia, heart block, ventricular arrhythmia), long QT syndrome, or current treatment with Class IA or Class III antiarrhythmic medicinal products.
* The participant had tested positive for the human immunodeficiency virus antibody, hepatitis C antibody, or hepatitis B surface antigen.
* The participant had a history of cancer within 6 months of enrolment, with the exception of basal cell carcinoma.
* Participant was a CYP2D6 IM, EM or URM and was taking a strong or moderate CYP2D6 inhibitor concomitantly with a strong or moderate CYP3A inhibitor.
* Participant was a CYP2D6 PM having taken a strong CYP3A inhibitor within 2 weeks prior to enrolment.
* If a female participant of childbearing potential had a positive pregnancy test (blood β-human chorionic gonadotropin [β-HCG]) or was breastfeeding prior to first dosing of eliglustat in this study, the participant could not enroll in the study at that time, but might have been rescreened after the end of the pregnancy, and/or when she was no longer breast feeding, provided rescreening took place before the end of the enrollment period.
* Women of childbearing potential who were unwilling or unable to be tested for pregnancy.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Investigational Site Number 124002, Montreal, Canada
- Russia (2):
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643002, Saint Petersburg
- Investigational Site Number 788001, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 active sites in 3 countries. A total of 33 participants were screened between 27 October 2015 and 07 June 2017, of which 2 participants were screen failures as the selection criteria were not met.
Pre-assignment Details: A total of 31 participants who completed one of the Phase 2 (GZGD00304 [NCT00358150]) or Phase 3 studies (GZGD02507 [ENGAGE; NCT00891202], GZGD02607 [ENCORE; NCT00943111], or GZGD03109 [EDGE; NCT01074944]) were enrolled in this current study (EFC13781) considered as an extension of these previous studies, and received treatment with eliglustat in the current (EFC13781) study.
Period: Overall Study
Arm/Group | Eliglustat
Started | 31
Completed | 27
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the full analysis set (FAS) population defined as all participants enrolled who received at least 1 dose of eliglustat treatment in the current study.
Groups:
- Eliglustat: Participants who completed one of the Phase 2 (GZGD00304) or Phase 3 studies (GZGD02507, GZGD02607 or GZGD03109) were enrolled in this current (EFC13781) study. Participants who were CYP2D6 IM, EM and URM received eliglustat 84 mg twice daily and participants who were CYP2D6 PM received eliglustat 84 mg once daily, for duration of minimum 2 years (unless early discontinuation occurred) and up to 4 years, or until commercial eliglustat was available to participants through reimbursement or through the compassionate use (expanded access) program.
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Age provided in this baseline measure defines the participant age at first dose of Eliglustat in the current study EFC13781 (in years).
  years | 36.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Time since first symptom of Gaucher to enrollment in EFC13781 [Mean (Standard Deviation); unit: years] | 22.6 (11.0)
Time since initial Gaucher diagnosis to enrollment in EFC13781 [Mean (Standard Deviation); unit: years] | 15.8 (9.2)
CYP2D6 metabolizer status [Count of Participants; unit: Participants] — Data represents participants who were CYP2D6 intermediate metabolizer (IM), extensive metabolizer (EM), poor metabolizer (PM) and ultra-rapid metabolizers (URM) at the Baseline.
  Participants
    CYP2D6 EM | 28
    CYP2D6 IM | 1
    CYP2D6 PM | 1
    CYP2D6 URM | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mobility Status Assessments at Study Baseline, Weeks 52, 104, 156 and 208
Description: Mobility, i.e., ability to walk was assessed as a part of Gaucher disease assessment in participants. In this outcome measure, number of participants with their different mobility status along with the use of mobility aids (unrestricted mobility, walks with difficulty, walks with orthopaedic aid, requires wheelchair, bedridden) at specified time points were reported. Baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: Analysis was performed on FAS population. Here, "number analyzed" = participants with available data for each specified category. Baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
Participants
  Unrestricted mobility: Study Baseline | 31
  Walks with difficulty: Study Baseline | 0
  Walks with orthopedic aid: Study Baseline | 0
  Requires wheelchair: Study Baseline | 0
  Bedridden: Study Baseline | 0
  Unrestricted mobility: Week 52 | 31
  Walks with difficulty: Week 52 | 0
  Walks with orthopedic aid: Week 52 | 0
  Requires wheelchair: Week 52 | 0
  Bedridden: Week 52 | 0
  Unrestricted mobility: Week 104: number analyzed (Participants) | 29
  Unrestricted mobility: Week 104 | 28
  Walks with Difficulty: Week 104: number analyzed (Participants) | 29
  Walks with Difficulty: Week 104 | 1
  Walks with orthopedic aid: Week 104: number analyzed (Participants) | 29
  Walks with orthopedic aid: Week 104 | 0
  Requires wheelchair: Week 104: number analyzed (Participants) | 29
  Requires wheelchair: Week 104 | 0
  Bedridden: Week 104: number analyzed (Participants) | 29
  Bedridden: Week 104 | 0
  Unrestricted mobility: Week 156: number analyzed (Participants) | 29
  Unrestricted mobility: Week 156 | 29
  Walks with difficulty: Week 156: number analyzed (Participants) | 29
  Walks with difficulty: Week 156 | 0
  Walks with orthopedic aid: Week 156: number analyzed (Participants) | 29
  Walks with orthopedic aid: Week 156 | 0
  Requires wheelchair: Week 156: number analyzed (Participants) | 29
  Requires wheelchair: Week 156 | 0
  Bedridden: Week 156: number analyzed (Participants) | 29
  Bedridden: Week 156 | 0
  Unrestricted mobility: Week 208: number analyzed (Participants) | 29
  Unrestricted mobility: Week 208 | 29
  Walks with difficulty: Week 208: number analyzed (Participants) | 29
  Walks with difficulty: Week 208 | 0
  Walks with orthopedic aid: Week 208: number analyzed (Participants) | 29
  Walks with orthopedic aid: Week 208 | 0
  Requires wheelchair: Week 208: number analyzed (Participants) | 29
  Requires wheelchair: Week 208 | 0
  Bedridden: Week 208: number analyzed (Participants) | 29
  Bedridden: Week 208 | 0

2. Primary Outcome: Number of Participants With Bone Pain Levels During the Past 4 Weeks at Study Baseline, Weeks 52, 104, 156 and 208
Description: Bone pain was assessed as a part of Gaucher disease assessment in participants. Participants were categorized as none (no bone pain), very mild bone pain, mild bone pain, moderate bone pain, severe bone pain and extreme bone pain during the past 4 weeks at each specified visit. In this outcome measure, number of participants with different level of bone pain during the past 4 weeks at specified time points were reported. Baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
Participants
  None: Study Baseline | 28
  Very Mild: Study Baseline | 1
  Mild: Study Baseline | 1
  Moderate: Study Baseline | 1
  Severe: Study Baseline | 0
  Extreme: Study Baseline | 0
  None: Week 52 | 29
  Very Mild: Week 52 | 1
  Mild: Week 52 | 0
  Moderate: Week 52 | 1
  Severe: Week 52 | 0
  Extreme: Week 52 | 0
  None: Week 104: number analyzed (Participants) | 29
  None: Week 104 | 28
  Very Mild: Week 104: number analyzed (Participants) | 29
  Very Mild: Week 104 | 1
  Mild: Week 104: number analyzed (Participants) | 29
  Mild: Week 104 | 0
  Moderate: Week 104: number analyzed (Participants) | 29
  Moderate: Week 104 | 0
  Severe: Week 104: number analyzed (Participants) | 29
  Severe: Week 104 | 0
  Extreme: Week 104: number analyzed (Participants) | 29
  Extreme: Week 104 | 0
  None: Week 156: number analyzed (Participants) | 29
  None: Week 156 | 29
  Very mild: Week 156: number analyzed (Participants) | 29
  Very mild: Week 156 | 0
  Mild: Week 156: number analyzed (Participants) | 29
  Mild: Week 156 | 0
  Moderate: Week 156: number analyzed (Participants) | 29
  Moderate: Week 156 | 0
  Severe: Week 156: number analyzed (Participants) | 29
  Severe: Week 156 | 0
  Extreme: Week 156: number analyzed (Participants) | 29
  Extreme: Week 156 | 0
  None: Week 208: number analyzed (Participants) | 29
  None: Week 208 | 28
  Very Mild: Week 208: number analyzed (Participants) | 29
  Very Mild: Week 208 | 1
  Mild: Week 208: number analyzed (Participants) | 29
  Mild: Week 208 | 0
  Moderate: Week 208: number analyzed (Participants) | 29
  Moderate: Week 208 | 0
  Severe: Week 208: number analyzed (Participants) | 29
  Severe: Week 208 | 0
  Extreme: Week 208: number analyzed (Participants) | 29
  Extreme: Week 208 | 0

3. Primary Outcome: Number of Participants With Bone Crisis at Study Baseline, Weeks 52, 104, 156 and 208
Description: Bone crisis was assessed as a part of Gaucher disease assessment in participants. Acute, excruciating episodic bone pain is characteristic of Gaucher bone crisis, which typically causes periosteal elevation, elevated white blood cell count, fever, or debilitation lasting several days or longer and requires treatment with immobilization of the affected area, and opioid analgesics. Participants were categorized as 0= no bone crisis, 1= 1 bone crisis, 2= 2 bone crisis and >=3 = more than 3 bone crisis during the assessment period. In this outcome measure, number of participants with different bone crises levels at specified time points were reported. Baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
Participants
  Bone Crisis (0): Study Baseline | 31
  Bone Crisis (1): Study Baseline | 0
  Bone Crisis (2): Study Baseline | 0
  Bone Crisis (>=3): Study Baseline | 0
  Bone Crisis (0): Week 52 | 31
  Bone Crisis (1): Week 52 | 0
  Bone Crisis (2): Week 52 | 0
  Bone Crisis (>=3): Week 52 | 0
  Bone Crisis (0): Week 104: number analyzed (Participants) | 29
  Bone Crisis (0): Week 104 | 29
  Bone Crisis (1): Week 104: number analyzed (Participants) | 29
  Bone Crisis (1): Week 104 | 0
  Bone Crisis (2): Week 104: number analyzed (Participants) | 29
  Bone Crisis (2): Week 104 | 0
  Bone Crisis (>=3): Week 104: number analyzed (Participants) | 29
  Bone Crisis (>=3): Week 104 | 0
  Bone Crisis (0): Week 156: number analyzed (Participants) | 29
  Bone Crisis (0): Week 156 | 28
  Bone Crisis (1): Week 156: number analyzed (Participants) | 29
  Bone Crisis (1): Week 156 | 1
  Bone Crisis (2): Week 156: number analyzed (Participants) | 29
  Bone Crisis (2): Week 156 | 0
  Bone Crisis (>=3): Week 156: number analyzed (Participants) | 29
  Bone Crisis (>=3): Week 156 | 0
  Bone Crisis (0): Week 208: number analyzed (Participants) | 29
  Bone Crisis (0): Week 208 | 29
  Bone Crisis (1): Week 208: number analyzed (Participants) | 29
  Bone Crisis (1): Week 208 | 0
  Bone Crisis (2): Week 208: number analyzed (Participants) | 29
  Bone Crisis (2): Week 208 | 0
  Bone Crisis (>=3): Week 208: number analyzed (Participants) | 29
  Bone Crisis (>=3): Week 208 | 0

4. Primary Outcome: Change From Current Study Baseline in Total Bone Marrow Burden (BMB) Scores at Weeks 52, 104, 156 and 208
Description: Bone marrow burden (BMB) scores indicate the degree of bone marrow infiltration. BMB score was measured using MRI (magnetic resonance imaging (MRI), ranged from 0 (no abnormalities) to 8 points (severe disease) for the lumbar spine and from 0 (no abnormalities) to 8 points (severe disease) for the femurs. The total BMB score was calculated as the sum of scores for femur and lumbar spine regions which ranged from 0 (no abnormalities) to 16 (severe disease) points. A higher BMB score signified more severe bone marrow involvement. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
score on a scale
  Total BMB Score: Study Baseline: number analyzed (Participants) | 28
  Total BMB Score: Study Baseline | 8.6667 (3.3860)
  Total BMB Score: Week 52: number analyzed (Participants) | 29
  Total BMB Score: Week 52 | 8.5057 (2.6482)
  Total BMB Score: Change at Week 52: number analyzed (Participants) | 26
  Total BMB Score: Change at Week 52 | -0.0256 (1.6969)
  Total BMB Score: Week 104: number analyzed (Participants) | 27
  Total BMB Score: Week 104 | 9.1111 (2.9627)
  Total BMB Score: Change at Week 104: number analyzed (Participants) | 24
  Total BMB Score: Change at Week 104 | 1.2639 (2.0897)
  Total BMB Score: Week 156: number analyzed (Participants) | 26
  Total BMB Score: Week 156 | 8.7821 (2.6178)
  Total BMB Score: Change at Week 156: number analyzed (Participants) | 23
  Total BMB Score: Change at Week 156 | 0.7101 (1.8404)
  Total BMB Score: Week 208: number analyzed (Participants) | 25
  Total BMB Score: Week 208 | 8.9067 (2.8844)
  Total BMB Score: Change at Week 208: number analyzed (Participants) | 22
  Total BMB Score: Change at Week 208 | 0.8939 (2.4023)

5. Primary Outcome: Change From Eliglustat Baseline in Total Bone Marrow Burden (BMB) Scores at Weeks 52, 104, 156 and 208
Description: Bone marrow burden (BMB) scores indicate the degree of bone marrow infiltration was measured using MRI, ranged from 0 (no abnormalities) to 8 points (severe disease) for the lumbar spine and from 0 (no abnormalities) to 8 points (severe disease) for the femurs. The total BMB score was calculated as the sum of scores for femur and lumbar spine regions which ranged from 0 (no abnormalities) to 16 (severe disease) points. A higher BMB score signified more severe bone marrow involvement. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 52, 104, 156 and 208 of the current study
Population: Analysis was performed on FAS population. Here, "number analyzed" = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from Enzyme Replacement Therapy [ERT]).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Eliglustat: Participants From Phase 2, ENGAGE and EDGE: Participants who completed one of the Phase 2 (GZGD00304) or Phase 3 studies (GZGD02507 [ENGAGE], or GZGD03109 [EDGE]) were included in this current (EFC13781) study. Participants who were CYP2D6 IM, EM and URM received eliglustat 84 mg twice daily and participants who were CYP2D6 PM received eliglustat 84 mg once daily, for duration of minimum 2 years (unless early discontinuation occurred) and up to 4 years, or until commercial eliglustat was available to participants through reimbursement or through the compassionate use (expanded access) program.
- Eliglustat: Participants From ENCORE: Participants who completed study GZGD02607 (ENCORE) were included in this current (EFC13781) study. Participants who were CYP2D6 IM, EM and URM received eliglustat 84 mg twice daily and participants who were CYP2D6 PM received eliglustat 84 mg once daily, for duration of minimum 2 years (unless early discontinuation occurred) and up to 4 years, or until commercial eliglustat was available to participants through reimbursement or through the compassionate use (expanded access) program.
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 4
score on a scale
  Total BMB Score: Eliglustat Baseline: number analyzed (Participants) | 14 | 4
  Total BMB Score: Eliglustat Baseline | 10.4286 (2.8146) | 6.8333 (2.4114)
  Total BMB Score: Week 52: number analyzed (Participants) | 25 | 4
  Total BMB Score: Week 52 | 8.4533 (2.7502) | 8.8333 (2.1858)
  Total BMB Score: Change at Week 52: number analyzed (Participants) | 13 | 4
  Total BMB Score: Change at Week 52 | -1.7179 (2.0765) | 2.0000 (1.2472)
  Total BMB Score: Week 104: number analyzed (Participants) | 23 | 4
  Total BMB Score: Week 104 | 8.9420 (3.1537) | 10.0833 (1.2874)
  Total BMB Score: Change at Week 104: number analyzed (Participants) | 11 | 4
  Total BMB Score: Change at Week 104 | -0.1818 (2.0459) | 3.2500 (2.6580)
  Total BMB Score: Week 156: number analyzed (Participants) | 24 | 2
  Total BMB Score: Week 156 | 8.6250 (2.6600) | 10.6667 (0.9428)
  Total BMB Score: Change at Week 156: number analyzed (Participants) | 11 | 2
  Total BMB Score: Change at Week 156 | -1.2424 (2.3098) | 3.3333 (2.3570)
  Total BMB Score: Week 208: number analyzed (Participants) | 22 | 3
  Total BMB Score: Week 208 | 8.7879 (3.0334) | 9.7778 (1.3878)
  Total BMB Score: Change at Week 208: number analyzed (Participants) | 11 | 3
  Total BMB Score: Change at Week 208 | -1.0606 (2.7641) | 3.3333 (3.3830)

6. Primary Outcome: Change From Current Study Baseline in Total Spine and Femur Bone Mineral Density (BMD) at Weeks 52, 104, 156 and 208
Description: Bone Mineral Density (BMD) measurements of the spine and bilateral femur were acquired by dual energy X-Ray absorptiometry (DXA) scan. Worst total femur at Baseline refers to the "worst" diseased left or right femur at Baseline. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams per centimeter square (g/cm^2)
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
grams per centimeter square (g/cm^2)
  Total Spine BMD: Study Baseline | 1.1449 (0.1236)
  Total Spine BMD: Week 52: number analyzed (Participants) | 26
  Total Spine BMD: Week 52 | 1.1476 (0.1255)
  Total Spine BMD: Change at Week 52: number analyzed (Participants) | 26
  Total Spine BMD: Change at Week 52 | -0.0029 (0.0282)
  Total Spine BMD: Week 104: number analyzed (Participants) | 29
  Total Spine BMD: Week 104 | 1.1326 (0.1217)
  Total Spine BMD: Change at Week 104: number analyzed (Participants) | 29
  Total Spine BMD: Change at Week 104 | -0.0055 (0.0333)
  Total Spine BMD: Week 156: number analyzed (Participants) | 29
  Total Spine BMD: Week 156 | 1.1373 (0.1173)
  Total Spine BMD: Change at Week 156: number analyzed (Participants) | 29
  Total Spine BMD: Change at Week 156 | -0.0007 (0.0484)
  Total Spine BMD: Week 208: number analyzed (Participants) | 26
  Total Spine BMD: Week 208 | 1.1236 (0.1146)
  Total Spine BMD: Change at Week 208: number analyzed (Participants) | 26
  Total Spine BMD: Change at Week 208 | -0.0120 (0.0550)
  Worst Total Femur BMD: Study Baseline | 1.0567 (0.1449)
  Worst Total Femur BMD: Week 52: number analyzed (Participants) | 26
  Worst Total Femur BMD: Week 52 | 1.0538 (0.1423)
  Worst Total Femur BMD: Change at Week 52: number analyzed (Participants) | 26
  Worst Total Femur BMD: Change at Week 52 | 0.0035 (0.0188)
  Worst Total Femur BMD: Week 104: number analyzed (Participants) | 29
  Worst Total Femur BMD: Week 104 | 1.0416 (0.1394)
  Worst Total Femur BMD: Change at Week 104: number analyzed (Participants) | 29
  Worst Total Femur BMD: Change at Week 104 | -0.0030 (0.0222)
  Worst Total Femur BMD: Week 156: number analyzed (Participants) | 28
  Worst Total Femur BMD: Week 156 | 1.0437 (0.1411)
  Worst Total Femur BMD: Change at Week 156: number analyzed (Participants) | 28
  Worst Total Femur BMD: Change at Week 156 | 0.0021 (0.0364)
  Worst Total Femur BMD: Week 208: number analyzed (Participants) | 26
  Worst Total Femur BMD: Week 208 | 1.0412 (0.1465)
  Worst Total Femur BMD: Change at Week 208: number analyzed (Participants) | 26
  Worst Total Femur BMD: Change at Week 208 | -0.0015 (0.0560)

7. Primary Outcome: Change From Eliglustat Baseline in Total Spine and Femur Bone Mineral Density (BMD) at Weeks 52, 104, 156 and 208
Description: BMD measurements of the spine and bilateral femur were acquired by DXA scan. Worst total femur at Baseline refers to the "worst" diseased left or right femur at baseline. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 52, 104, 156 and 208 of the current study
Population: Analysis was performed on FAS population. Here, "number analyzed" = participants with available data for each specified category. Data for this outcome measure was was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 4
g/cm^2
  Total Spine BMD: Eliglustat Baseline: number analyzed (Participants) | 23 | 4
  Total Spine BMD: Eliglustat Baseline | 1.0757 (0.1322) | 1.1350 (0.0896)
  Total Spine BMD: Week 52: number analyzed (Participants) | 24 | 2
  Total Spine BMD: Week 52 | 1.1495 (0.1307) | 1.1245 (0.0035)
  Total Spine BMD: Change at Week 52: number analyzed (Participants) | 20 | 2
  Total Spine BMD: Change at Week 52 | 0.0582 (0.0656) | 0.0195 (0.0530)
  Total Spine BMD: Week 104: number analyzed (Participants) | 25 | 4
  Total Spine BMD: Week 104 | 1.1280 (0.1216) | 1.1615 (0.1371)
  Total Spine BMD: Change at Week 104: number analyzed (Participants) | 21 | 4
  Total Spine BMD: Change at Week 104 | 0.0600 (0.0633) | 0.0265 (0.0617)
  Total Spine BMD: Week 156: number analyzed (Participants) | 25 | 4
  Total Spine BMD: Week 156 | 1.1354 (0.1153) | 1.1498 (0.1480)
  Total Spine BMD: Change at Week 156: number analyzed (Participants) | 21 | 4
  Total Spine BMD: Change at Week 156 | 0.0712 (0.0718) | 0.0148 (0.0692)
  Total Spine BMD: Week 208: number analyzed (Participants) | 23 | 3
  Total Spine BMD: Week 208 | 1.1168 (0.1120) | 1.1757 (0.1466)
  Total Spine BMD: Change at Week 208: number analyzed (Participants) | 19 | 3
  Total Spine BMD: Change at Week 208 | 0.0616 (0.0799) | 0.0190 (0.0596)
  Worst Total Femur BMD: Eliglustat Baseline: number analyzed (Participants) | 23 | 4
  Worst Total Femur BMD: Eliglustat Baseline | 1.0330 (0.1550) | 1.1600 (0.1356)
  Worst Total Femur BMD: Week 52: number analyzed (Participants) | 20 | 3
  Worst Total Femur BMD: Week 52 | 1.0643 (0.1565) | 1.0853 (0.0634)
  Worst Total Femur BMD: Change at Week 52: number analyzed (Participants) | 20 | 3
  Worst Total Femur BMD: Change at Week 52 | 0.0169 (0.0495) | -0.0080 (0.0686)
  Worst Total Femur BMD: Week 104: number analyzed (Participants) | 21 | 4
  Worst Total Femur BMD: Week 104 | 1.0346 (0.1485) | 1.1260 (0.1253)
  Worst Total Femur BMD: Change at Week 104: number analyzed (Participants) | 21 | 4
  Worst Total Femur BMD: Change at Week 104 | 0.0118 (0.0460) | -0.0340 (0.0551)
  Worst Total Femur BMD: Week 156: number analyzed (Participants) | 21 | 4
  Worst Total Femur BMD: Week 156 | 1.0380 (0.1515) | 1.1328 (0.1358)
  Worst Total Femur BMD: Change at Week 156: number analyzed (Participants) | 21 | 4
  Worst Total Femur BMD: Change at Week 156 | 0.0152 (0.0586) | -0.0273 (0.0614)
  Worst Total Femur BMD: Week 208: number analyzed (Participants) | 19 | 3
  Worst Total Femur BMD: Week 208 | 1.0304 (0.1547) | 1.1430 (0.1572)
  Worst Total Femur BMD: Change at Week 208: number analyzed (Participants) | 19 | 3
  Worst Total Femur BMD: Change at Week 208 | 0.0198 (0.0598) | -0.0503 (0.0715)

8. Primary Outcome: Change From Current Study Baseline in Spine and Femur Total T-Scores for BMD at Weeks 52, 104, 156 and 208
Description: BMD measurements of the spine and bilateral femur were acquired by DXA scan. The T-score bone density categories were: normal (score >-1), osteopenia (score -2.5 to <=-1), and osteoporosis (score <= -2.5). Worst total femur at Baseline refers to the "worst" diseased left or right femur at baseline. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
T-score
  Total Spine T-score: Study Baseline | -0.4413 (0.9782)
  Total Spine T-score: Week 52: number analyzed (Participants) | 26
  Total Spine T-score: Week 52 | -0.4362 (1.0155)
  Total Spine T-score: Change at Week 52: number analyzed (Participants) | 26
  Total Spine T-score: Change at Week 52 | -0.0250 (0.2356)
  Total Spine T-score: Week 104: number analyzed (Participants) | 29
  Total Spine T-score: Week 104 | -0.5566 (0.9522)
  Total Spine T-score: Change at Week 104: number analyzed (Participants) | 29
  Total Spine T-score: Change at Week 104 | -0.0479 (0.2751)
  Total Spine T-score: Week 156: number analyzed (Participants) | 29
  Total Spine T-score: Week 156 | -0.5152 (0.9075)
  Total Spine T-score: Change at Week 156: number analyzed (Participants) | 29
  Total Spine T-score: Change at Week 156 | -0.0066 (0.4013)
  Total Spine T-score: Week 208: number analyzed (Participants) | 26
  Total Spine T-score: Week 208 | -0.6238 (0.9015)
  Total Spine T-score: Change at Week 208: number analyzed (Participants) | 26
  Total Spine T-score: Change at Week 208 | -0.1012 (0.4580)
  Worst Total Femur T-score: Study Baseline | 0.0119 (1.0001)
  Worst Total Femur T-score: Week 52: number analyzed (Participants) | 26
  Worst Total Femur T-score: Week 52 | -0.0119 (1.0104)
  Worst Total Femur T-score: Change at Week 52: number analyzed (Participants) | 26
  Worst Total Femur T-score: Change at Week 52 | 0.0273 (0.1481)
  Worst Total Femur T-score: Week 104: number analyzed (Participants) | 29
  Worst Total Femur T-score: Week 104 | -0.1345 (0.8867)
  Worst Total Femur T-score: Change at Week 104: number analyzed (Participants) | 29
  Worst Total Femur T-score: Change at Week 104 | -0.0245 (0.1670)
  Worst Total Femur T-score: Week 156: number analyzed (Participants) | 28
  Worst Total Femur T-score: Week 156 | -0.1032 (0.9087)
  Worst Total Femur T-score: Change at Week 156: number analyzed (Participants) | 28
  Worst Total Femur T-score: Change at Week 156 | 0.0179 (0.2704)
  Worst Total Femur T-score: Week 208: number analyzed (Participants) | 26
  Worst Total Femur T-score: Week 208 | -0.1196 (0.9594)
  Worst Total Femur T-score: Change at Week 208: number analyzed (Participants) | 26
  Worst Total Femur T-score: Change at Week 208 | -0.0073 (0.4318)

9. Primary Outcome: Change From Eliglustat Baseline in Spine and Femur Total T-Scores for BMD at Weeks 52, 104, 156 and 208
Description: BMD measurements of the spine and bilateral femur were acquired by DXA scan. The T-score bone density categories were: normal (score >-1), osteopenia (score -2.5 to <=-1), and osteoporosis (score <= -2.5). Worst total femur at Baseline refers to the "worst" diseased left or right femur at baseline. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 52, 104, 156 and 208 of the current study
Population: Analysis was performed on FAS population. Here, "number analyzed" = participants with available data for each specified category. Here, "0" signifies that none of the participants were available for assessment at the specified timepoint. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 4
T-score
  Total Spine T-score: Eliglustat Baseline: number analyzed (Participants) | 21 | 2
  Total Spine T-score: Eliglustat Baseline | -0.9381 (1.0443) | -0.3000 (0.8485)
  Total Spine T-score: Week 52: number analyzed (Participants) | 24 | 2
  Total Spine T-score: Week 52 | -0.4063 (1.0530) | -0.7950 (0.0354)
  Total Spine T-score: Change at Week 52: number analyzed (Participants) | 19 | 0
  Total Spine T-score: Change at Week 52 | 0.5126 (0.5622) |
  Total Spine T-score: Week 104: number analyzed (Participants) | 25 | 4
  Total Spine T-score: Week 104 | -0.5808 (0.9512) | -0.4050 (1.0898)
  Total Spine T-score: Change at Week 104: number analyzed (Participants) | 20 | 2
  Total Spine T-score: Change at Week 104 | 0.5215 (0.5229) | 0.5200 (0.5657)
  Total Spine T-score: Week 156: number analyzed (Participants) | 25 | 4
  Total Spine T-score: Week 156 | -0.5172 (0.8875) | -0.5025 (1.1771)
  Total Spine T-score: Change at Week 156: number analyzed (Participants) | 20 | 2
  Total Spine T-score: Change at Week 156 | 0.6150 (0.6000) | 0.4300 (0.7495)
  Total Spine T-score: Week 208: number analyzed (Participants) | 23 | 3
  Total Spine T-score: Week 208 | -0.6570 (0.8823) | -0.3700 (1.2194)
  Total Spine T-score: Change at Week 208: number analyzed (Participants) | 18 | 1
  Total Spine T-score: Change at Week 208 | 0.5544 (0.6867) | 0.7300
  Worst Total Femur T-score: Eliglustat Baseline: number analyzed (Participants) | 21 | 2
  Worst Total Femur T-score: Eliglustat Baseline | -0.0190 (1.0939) | 1.1000 (0.9899)
  Worst Total Femur T-score: Week 52: number analyzed (Participants) | 19 | 1
  Worst Total Femur T-score: Week 52 | 0.1142 (1.1458) | 0.3800
  Worst Total Femur T-score: Change at Week 52: number analyzed (Participants) | 19 | 1
  Worst Total Femur T-score: Change at Week 52 | 0.0616 (0.3755) | -0.0200
  Worst Total Femur T-score: Week 104: number analyzed (Participants) | 20 | 2
  Worst Total Femur T-score: Week 104 | -0.0950 (0.9778) | 0.8200 (0.6647)
  Worst Total Femur T-score: Change at Week 104: number analyzed (Participants) | 20 | 2
  Worst Total Femur T-score: Change at Week 104 | 0.0400 (0.3661) | -0.2800 (0.3253)
  Worst Total Femur T-score: Week 156: number analyzed (Participants) | 20 | 2
  Worst Total Femur T-score: Week 156 | -0.0615 (1.0000) | 0.9050 (0.7283)
  Worst Total Femur T-score: Change at Week 156: number analyzed (Participants) | 20 | 2
  Worst Total Femur T-score: Change at Week 156 | 0.0735 (0.4602) | -0.1950 (0.2616)
  Worst Total Femur T-score: Week 208: number analyzed (Participants) | 18 | 1
  Worst Total Femur T-score: Week 208 | -0.0867 (1.0293) | 1.3500
  Worst Total Femur T-score: Change at Week 208: number analyzed (Participants) | 18 | 1
  Worst Total Femur T-score: Change at Week 208 | 0.1022 (0.4355) | -0.4500

10. Primary Outcome: Change From Current Study Baseline in Spine and Femur Total Z-Scores for BMD at Weeks 52, 104, 156 and 208
Description: BMD measurements of the spine and bilateral femur were acquired by DXA scan. The Z-score bone density categories were: normal (score >-2) and below normal (score <=-2). Worst total femur at Baseline refers to the "worst" diseased left or right femur at baseline. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
Z-score
  Total Spine Z-score: Study Baseline | -0.3687 (0.8529)
  Total Spine Z-score: Week 52: number analyzed (Participants) | 26
  Total Spine Z-score: Week 52 | -0.3338 (0.8597)
  Total Spine Z-score: Change at Week 52: number analyzed (Participants) | 26
  Total Spine Z-score: Change at Week 52 | -0.0092 (0.2405)
  Total Spine Z-score: Week 104: number analyzed (Participants) | 29
  Total Spine Z-score: Week 104 | -0.4555 (0.8522)
  Total Spine Z-score: Change at Week 104: number analyzed (Participants) | 29
  Total Spine Z-score: Change at Week 104 | -0.0245 (0.2945)
  Total Spine Z-score: Week 156: number analyzed (Participants) | 29
  Total Spine Z-score: Week 156 | -0.4034 (0.8464)
  Total Spine Z-score: Change at Week 156: number analyzed (Participants) | 29
  Total Spine Z-score: Change at Week 156 | 0.0276 (0.4275)
  Total Spine Z-score: Week 208: number analyzed (Participants) | 26
  Total Spine Z-score: Week 208 | -0.5035 (0.8289)
  Total Spine Z-score: Change at Week 208: number analyzed (Participants) | 26
  Total Spine Z-score: Change at Week 208 | -0.0519 (0.4759)
  Worst Total Femur Z-score: Study Baseline | 0.1935 (0.9392)
  Worst Total Femur Z-score: Week 52: number analyzed (Participants) | 26
  Worst Total Femur Z-score: Week 52 | 0.2196 (0.9469)
  Worst Total Femur Z-score: Change at Week 52: number analyzed (Participants) | 26
  Worst Total Femur Z-score: Change at Week 52 | 0.0504 (0.1495)
  Worst Total Femur Z-score: Week 104: number analyzed (Participants) | 29
  Worst Total Femur Z-score: Week 104 | 0.0921 (0.8288)
  Worst Total Femur Z-score: Change at Week 104: number analyzed (Participants) | 29
  Worst Total Femur Z-score: Change at Week 104 | 0.0114 (0.1663)
  Worst Total Femur Z-score: Week 156: number analyzed (Participants) | 28
  Worst Total Femur Z-score: Week 156 | 0.1521 (0.8500)
  Worst Total Femur Z-score: Change at Week 156: number analyzed (Participants) | 28
  Worst Total Femur Z-score: Change at Week 156 | 0.0757 (0.2705)
  Worst Total Femur Z-score: Week 208: number analyzed (Participants) | 26
  Worst Total Femur Z-score: Week 208 | 0.1408 (0.9077)
  Worst Total Femur Z-score: Change at Week 208: number analyzed (Participants) | 26
  Worst Total Femur Z-score: Change at Week 208 | 0.0746 (0.4267)

11. Primary Outcome: Change From Eliglustat Baseline in Spine and Femur Total Z-Scores for BMD at Weeks 52, 104, 156 and 208
Description: BMD measurements of the spine and bilateral femur were acquired by DXA scan. The Z-score bone density categories are: normal (score >-2) and below normal (score <=-2). Worst total femur at Baseline refers to the "worst" diseased left or right femur at baseline. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 52, 104, 156 and 208 of the current study
Population: Analysis was performed on FAS population. Here, "number analyzed" = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 4
Z-score
  Total Spine Z-score: Eliglustat Baseline: number analyzed (Participants) | 23 | 4
  Total Spine Z-score: Eliglustat Baseline | -0.8826 (0.9824) | -0.5750 (0.6185)
  Total Spine Z-score: Week 52: number analyzed (Participants) | 24 | 2
  Total Spine Z-score: Week 52 | -0.2954 (0.8851) | -0.7950 (0.0354)
  Total Spine Z-score: Change at Week 52: number analyzed (Participants) | 20 | 2
  Total Spine Z-score: Change at Week 52 | 0.5030 (0.4230) | 0.0550 (0.3889)
  Total Spine Z-score: Week 104: number analyzed (Participants) | 25 | 4
  Total Spine Z-score: Week 104 | -0.4636 (0.8357) | -0.4050 (1.0898)
  Total Spine Z-score: Change at Week 104: number analyzed (Participants) | 21 | 4
  Total Spine Z-score: Change at Week 104 | 0.5186 (0.4578) | 0.1700 (0.5553)
  Total Spine Z-score: Week 156: number analyzed (Participants) | 25 | 4
  Total Spine Z-score: Week 156 | -0.3876 (0.8129) | -0.5025 (1.1771)
  Total Spine Z-score: Change at Week 156: number analyzed (Participants) | 21 | 4
  Total Spine Z-score: Change at Week 156 | 0.6276 (0.5671) | 0.0725 (0.6233)
  Total Spine Z-score: Week 208: number analyzed (Participants) | 23 | 3
  Total Spine Z-score: Week 208 | -0.5209 (0.8017) | -0.3700 (1.2194)
  Total Spine Z-score: Change at Week 208: number analyzed (Participants) | 19 | 3
  Total Spine Z-score: Change at Week 208 | 0.5716 (0.6454) | 0.0967 (0.5615)
  Worst Total Femur Z-score: Eliglustat Baseline: number analyzed (Participants) | 23 | 4
  Worst Total Femur Z-score: Eliglustat Baseline | 0.0826 (1.0373) | 0.5000 (0.8287)
  Worst Total Femur Z-score: Week 52: number analyzed (Participants) | 20 | 3
  Worst Total Femur Z-score: Week 52 | 0.3475 (1.0593) | 0.1100 (0.5071)
  Worst Total Femur Z-score: Change at Week 52: number analyzed (Participants) | 20 | 3
  Worst Total Femur Z-score: Change at Week 52 | 0.1825 (0.3842) | 0.0100 (0.4530)
  Worst Total Femur Z-score: Week 104: number analyzed (Participants) | 21 | 4
  Worst Total Femur Z-score: Week 104 | 0.1429 (0.9361) | 0.3375 (0.7968)
  Worst Total Femur Z-score: Change at Week 104: number analyzed (Participants) | 21 | 4
  Worst Total Femur Z-score: Change at Week 104 | 0.1571 (0.3503) | -0.1625 (0.3728)
  Worst Total Femur Z-score: Week 156: number analyzed (Participants) | 21 | 4
  Worst Total Femur Z-score: Week 156 | 0.1876 (0.9632) | 0.3975 (0.8695)
  Worst Total Femur Z-score: Change at Week 156: number analyzed (Participants) | 21 | 4
  Worst Total Femur Z-score: Change at Week 156 | 0.2019 (0.4407) | -0.1025 (0.4180)
  Worst Total Femur Z-score: Week 208: number analyzed (Participants) | 19 | 3
  Worst Total Femur Z-score: Week 208 | 0.1758 (0.9830) | 0.2700 (1.0789)
  Worst Total Femur Z-score: Change at Week 208: number analyzed (Participants) | 19 | 3
  Worst Total Femur Z-score: Change at Week 208 | 0.2495 (0.4439) | -0.2633 (0.4652)

12. Primary Outcome: Total Number of New or Worsening Osteonecrosis Events for Spine and Femur at Study Baseline, Week 52, 104, 156 and 208
Description: Osteonecrosis was assessed by bone MRI and X-Ray for spine and by MRI for femur. Total number of new or worsening osteonecrosis events among all the participants with corresponding assessment at specified time points were reported in this outcome measure. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Full Range); unit: events
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events
  Spine Osteonecrosis (MRI): Study Baseline: number analyzed (Participants) | 25
  Spine Osteonecrosis (MRI): Study Baseline | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (MRI): Week 52: number analyzed (Participants) | 29
  Spine Osteonecrosis (MRI): Week 52 | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (MRI): Week 104: number analyzed (Participants) | 27
  Spine Osteonecrosis (MRI): Week 104 | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (MRI): Week 156: number analyzed (Participants) | 26
  Spine Osteonecrosis (MRI): Week 156 | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (MRI): Week 208: number analyzed (Participants) | 24
  Spine Osteonecrosis (MRI): Week 208 | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (X-ray): Study Baseline: number analyzed (Participants) | 24
  Spine Osteonecrosis (X-ray): Study Baseline | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (X-ray): Week 104: number analyzed (Participants) | 27
  Spine Osteonecrosis (X-ray): Week 104 | 0.0000 [0.000 to 0.000]
  Spine Osteonecrosis (X-ray): Week 208: number analyzed (Participants) | 21
  Spine Osteonecrosis (X-ray): Week 208 | 0.0000 [0.000 to 0.000]
  Femur Osteonecrosis (MRI): Study Baseline: number analyzed (Participants) | 29
  Femur Osteonecrosis (MRI): Study Baseline | 0.0690 [0.000 to 1.000]
  Femur Osteonecrosis (MRI): Week 52: number analyzed (Participants) | 29
  Femur Osteonecrosis (MRI): Week 52 | 0.0345 [0.000 to 1.000]
  Femur Osteonecrosis (MRI): Week 104: number analyzed (Participants) | 28
  Femur Osteonecrosis (MRI): Week 104 | 0.0000 [0.000 to 0.000]
  Femur Osteonecrosis (MRI): Week 156: number analyzed (Participants) | 26
  Femur Osteonecrosis (MRI): Week 156 | 0.0385 [0.000 to 1.000]
  Femur Osteonecrosis (MRI): Week 208: number analyzed (Participants) | 24
  Femur Osteonecrosis (MRI): Week 208 | 0.0000 [0.000 to 0.000]

13. Primary Outcome: Total Number of New or Worsening Fracture Events for Spine and Femur at Study Baseline, Week 52, 104, 156 and 208
Description: Fracture was assessed by bone MRI and X-Ray for spine and by MRI for femur. Total number of new or worsening fracture events among all the participants with corresponding assessment at specified time points were reported in this outcome measure. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Full Range); unit: events
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events
  Spine Fracture (MRI): Study Baseline: number analyzed (Participants) | 25
  Spine Fracture (MRI): Study Baseline | 0.0000 [0.000 to 0.000]
  Spine Fracture (MRI): Week 52: number analyzed (Participants) | 29
  Spine Fracture (MRI): Week 52 | 0.0690 [0.000 to 2.000]
  Spine Fracture (MRI): Week 104: number analyzed (Participants) | 27
  Spine Fracture (MRI): Week 104 | 0.0000 [0.000 to 0.000]
  Spine Fracture (MRI): Week 156: number analyzed (Participants) | 26
  Spine Fracture (MRI): Week 156 | 0.0000 [0.000 to 0.000]
  Spine Fracture (MRI): Week 208: number analyzed (Participants) | 24
  Spine Fracture (MRI): Week 208 | 0.0417 [0.000 to 1.000]
  Spine Fracture (X-ray): Study Baseline: number analyzed (Participants) | 24
  Spine Fracture (X-ray): Study Baseline | 0.0000 [0.000 to 0.000]
  Spine Fracture (X-ray): Week 104: number analyzed (Participants) | 27
  Spine Fracture (X-ray): Week 104 | 0.0741 [0.000 to 2.000]
  Spine Fracture (X-ray): Week 208: number analyzed (Participants) | 21
  Spine Fracture (X-ray): Week 208 | 0.0000 [0.000 to 0.000]
  Femur Fracture (MRI): Study Baseline: number analyzed (Participants) | 29
  Femur Fracture (MRI): Study Baseline | 0.0000 [0.000 to 0.000]
  Femur Fracture (MRI): Week 52: number analyzed (Participants) | 29
  Femur Fracture (MRI): Week 52 | 0.0000 [0.000 to 0.000]
  Femur Fracture (MRI): Week 104: number analyzed (Participants) | 28
  Femur Fracture (MRI): Week 104 | 0.0000 [0.000 to 0.000]
  Femur Fracture (MRI): Week 156: number analyzed (Participants) | 26
  Femur Fracture (MRI): Week 156 | 0.0000 [0.000 to 0.000]
  Femur Fracture (MRI): Week 208: number analyzed (Participants) | 24
  Femur Fracture (MRI): Week 208 | 0.0000 [0.000 to 0.000]

14. Primary Outcome: Total Number of New or Worsening Infarcts Events for Spine and Femur at Study Baseline, Week 52, 104, 156 and 208
Description: Infarcts were assessed by bone MRI and X-Ray for spine and by MRI for femur. Total number of new or worsening infarcts events among all the participants with corresponding assessment at specified time points were reported in this outcome measure. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 52, 104, 156 and 208
Population: as for outcome 1
Measure: Mean (Full Range); unit: events
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events
  Spine Infarcts (MRI): Study Baseline: number analyzed (Participants) | 28
  Spine Infarcts (MRI): Study Baseline | 0.0000 [0.000 to 0.000]
  Spine Infarcts (MRI): Week 52: number analyzed (Participants) | 29
  Spine Infarcts (MRI): Week 52 | 0.0000 [0.000 to 0.000]
  Spine Infarcts (MRI): Week 104: number analyzed (Participants) | 27
  Spine Infarcts (MRI): Week 104 | 0.0000 [0.000 to 0.000]
  Spine Infarcts (MRI): Week 156: number analyzed (Participants) | 26
  Spine Infarcts (MRI): Week 156 | 0.0000 [0.000 to 0.000]
  Spine Infarcts (MRI): Week 208: number analyzed (Participants) | 24
  Spine Infarcts (MRI): Week 208 | 0.0000 [0.000 to 0.000]
  Spine Infarcts (X-ray): Study Baseline: number analyzed (Participants) | 26
  Spine Infarcts (X-ray): Study Baseline | 0.0000 [0.000 to 0.000]
  Spine Infarcts (X-ray): Week 104: number analyzed (Participants) | 27
  Spine Infarcts (X-ray): Week 104 | 0.0000 [0.000 to 0.000]
  Spine Infarcts (X-ray): Week 208: number analyzed (Participants) | 21
  Spine Infarcts (X-ray): Week 208 | 0.0000 [0.000 to 0.000]
  Femur Infarcts (MRI): Study Baseline: number analyzed (Participants) | 30
  Femur Infarcts (MRI): Study Baseline | 0.6000 [0.000 to 4.000]
  Femur Infarcts (MRI): Week 52: number analyzed (Participants) | 29
  Femur Infarcts (MRI): Week 52 | 0.2069 [0.000 to 2.000]
  Femur Infarcts (MRI): Week 104: number analyzed (Participants) | 28
  Femur Infarcts (MRI): Week 104 | 0.0000 [0.000 to 0.000]
  Femur Infarcts (MRI): Week 156: number analyzed (Participants) | 26
  Femur Infarcts (MRI): Week 156 | 0.0000 [0.000 to 0.000]
  Femur Infarcts (MRI): Week 208: number analyzed (Participants) | 24
  Femur Infarcts (MRI): Week 208 | 0.0417 [0.000 to 1.000]

15. Primary Outcome: Total Number of New or Worsening Lytic Lesions Events for Spine at Study Baseline, Week 104, and 208
Description: Lytic Lesions were assessed by bone X-Ray for spine. Total number of new or worsening lytic lesions events among all the participants with corresponding assessment at specified time points were reported in this outcome measure. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 104, and 208
Population: as for outcome 1
Measure: Mean (Full Range); unit: events
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events
  Spine Lytic Lesions (X-ray): Study Baseline: number analyzed (Participants) | 26
  Spine Lytic Lesions (X-ray): Study Baseline | 0.0385 [0.000 to 1.000]
  Spine Lytic Lesions (X-ray): Week 104: number analyzed (Participants) | 27
  Spine Lytic Lesions (X-ray): Week 104 | 0.0000 [0.000 to 0.000]
  Spine Lytic Lesions (X-ray): Week 208: number analyzed (Participants) | 21
  Spine Lytic Lesions (X-ray): Week 208 | 0.0000 [0.000 to 0.000]

16. Primary Outcome: Observed Annual Incidence Rate for Spine and Femur Osteonecrosis at Week 52, 104, 156 and 208
Description: Observed annual incidence rate was estimated using the total number of events divided by the total years of follow-up in each specified year (for all participants). Osteonecrosis was assessed by bone MRI and X-Ray for spine and by MRI for femur.
Time Frame: For 52 Weeks (i.e., 1 year),104 Weeks (i.e., 2 year), 156 Weeks (i.e., 3 year) and 208 Weeks (i.e., 4 years)
Population: Analysis was performed on FAS population.
Measure: Number; unit: events per participant-year
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events per participant-year
  Spine Osteonecrosis (MRI): Week 52 | 0
  Spine Osteonecrosis (MRI): Week 104 | 0
  Spine Osteonecrosis (MRI): Week 156 | 0
  Spine Osteonecrosis (MRI): Week 208 | 0
  Spine Osteonecrosis (X-ray): Week 104 | 0
  Spine Osteonecrosis (X-ray): Week 208 | 0
  Femur Osteonecrosis (MRI): Week 52 | 0.1013
  Femur Osteonecrosis (MRI): Week 104 | 0.0353
  Femur Osteonecrosis (MRI): Week 156 | 0.0384
  Femur Osteonecrosis (MRI): Week 208 | 0.0104

17. Primary Outcome: Observed Annual Incidence Rate for Spine and Femur Fracture at Week 52, 104, 156 and 208
Description: Observed annual incidence rate was estimated using the total number of events divided by the total years of follow-up in each specified year (for all participants). Fracture was assessed by bone MRI and X-Ray for spine and by MRI for femur.
Time Frame: For 52 Weeks (i.e., 1 year),104 Weeks (i.e., 2 year), 156 Weeks (i.e., 3 year) and 208 Weeks (i.e., 4 years)
Population: Analysis was performed on FAS population.
Measure: Number; unit: events per participant-year
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events per participant-year
  Spine Fracture (MRI): Week 52 | 0.1350
  Spine Fracture (MRI): Week 104 | 0.0366
  Spine Fracture(MRI): Week 156 | 0
  Spine Fracture (MRI): Week 208 | 0.0104
  Spine Fracture (X-ray): Week 104 | 0.0369
  Spine Fracture (X-ray): Week 208 | 0
  Femur Fracture (MRI): Week 52 | 0
  Femur Fracture (MRI): Week 104 | 0
  Femur Fracture (MRI): Week 156 | 0
  Femur Fracture (MRI): Week 208 | 0

18. Primary Outcome: Observed Annual Incidence Rate for Spine and Femur Infarcts at Week 52, 104, 156 and 208
Description: Observed annual incidence rate was estimated using the total number of events divided by the total years of follow-up in each specified year (for all participants). Infarcts were assessed by bone MRI and X-Ray for spine and by MRI for femur.
Time Frame: For 52 Weeks (i.e., 1 year),104 Weeks (i.e., 2 year), 156 Weeks (i.e., 3 year) and 208 Weeks (i.e., 4 years)
Population: Analysis was performed on FAS population.
Measure: Number; unit: events per participant-year
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events per participant-year
  Spine Infarcts (MRI): Week 52 | 0
  Spine Infarcts (MRI): Week 104 | 0
  Spine Infarcts (MRI): Week 156 | 0
  Spine Infarcts (MRI): Week 208 | 0
  Spine Infarcts (X-ray): Week 104 | 0
  Spine Infarcts (X-ray): Week 208 | 0
  Femur Infarcts (MRI): Week 52 | 0.6752
  Femur Infarcts (MRI): Week 104 | 0.2470
  Femur Infarcts (MRI): Week 156 | 0.1664
  Femur Infarcts (MRI): Week 208 | 0.1145

19. Primary Outcome: Observed Annual Incidence Rate for Spine Lytic Lesion at Week 104, and 208
Description: Observed annual incidence rate was estimated using the total number of events divided by the total years of follow-up in each specified year (for all participants). Lytic Lesions were assessed by bone X-Ray for spine.
Time Frame: For 104 Weeks (i.e., 2 year), and 208 Weeks (i.e., 4 years)
Population: Analysis was performed on FAS population.
Measure: Number; unit: events per participant-year
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
events per participant-year
  Spine Lytic Lesions (X-ray): Week 104 | 0
  Spine Lytic Lesions (X-ray): Week 208 | 0

20. Primary Outcome: Change From Current Study Baseline in Bone Biomarker Level: Macrophage Inflammatory Protein 1 Beta (MIP-1β) at Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Description: MIP-1β considered a biomarker of active bone disease, was assayed from plasma. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 26, 52, 78, 104, 130, 156, 182, 208 and 234
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
picograms per milliliter (pg/mL)
  Study Baseline: number analyzed (Participants) | 27
  Study Baseline | 175.8296 (114.6313)
  Change at Week 26: number analyzed (Participants) | 27
  Change at Week 26 | -36.0593 (78.2488)
  Change at Week 52: number analyzed (Participants) | 26
  Change at Week 52 | -31.4692 (97.6425)
  Change at Week 78: number analyzed (Participants) | 22
  Change at Week 78 | -16.6818 (93.2333)
  Change at Week 104: number analyzed (Participants) | 23
  Change at Week 104 | -33.0217 (77.0603)
  Change at Week 130: number analyzed (Participants) | 25
  Change at Week 130 | 897.1680 (4660.2892)
  Change at Week 156: number analyzed (Participants) | 25
  Change at Week 156 | 1008.8400 (5150.4257)
  Change at Week 182: number analyzed (Participants) | 25
  Change at Week 182 | 1007.9880 (5177.6248)
  Change at Week 208: number analyzed (Participants) | 23
  Change at Week 208 | 1381.6652 (6751.1152)
  Change at Week 234: number analyzed (Participants) | 9
  Change at Week 234 | 6721.9000 (20005.3684)

21. Primary Outcome: Change From Eliglustat Baseline in Bone Biomarker Level: Macrophage Inflammatory Protein 1 Beta (MIP-1β) at Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Description: MIP-1β considered a biomarker of active bone disease, was assayed from plasma. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234 of the current study
Population: Analyzed on FAS population. Here, "number analyzed" = participants with available data for each specified category and "0" in number analyzed field signifies that none of participants had evaluable data at specified timepoint. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 4
pg/mL
  Eliglustat Baseline: number analyzed (Participants) | 18 | 4
  Eliglustat Baseline | 265.3944 (149.3311) | 103.7750 (32.0705)
  Change at Week 26: number analyzed (Participants) | 18 | 4
  Change at Week 26 | -136.2167 (135.6276) | 66.7750 (70.3377)
  Change at Week 52: number analyzed (Participants) | 17 | 4
  Change at Week 52 | -153.7647 (127.0446) | 79.0750 (115.7302)
  Change at Week 78: number analyzed (Participants) | 14 | 4
  Change at Week 78 | -151.1857 (118.7980) | 37.7000 (79.6721)
  Change at Week 104: number analyzed (Participants) | 16 | 4
  Change at Week 104 | -152.8875 (128.7985) | 74.6750 (81.1326)
  Change at Week 130: number analyzed (Participants) | 16 | 4
  Change at Week 130 | -159.4750 (149.3802) | 53.6250 (86.1059)
  Change at Week 156: number analyzed (Participants) | 16 | 4
  Change at Week 156 | -141.7750 (129.3039) | 68.9000 (101.0239)
  Change at Week 182: number analyzed (Participants) | 16 | 4
  Change at Week 182 | -145.6750 (138.9781) | 46.6500 (64.9619)
  Change at Week 208: number analyzed (Participants) | 15 | 4
  Change at Week 208 | -149.8933 (153.1632) | 67.2500 (75.0664)
  Change at Week 234: number analyzed (Participants) | 7 | 0
  Change at Week 234 | -222.6857 (64.4851) |

22. Primary Outcome: Change From Current Study Baseline in Bone Biomarker Level: Procollagen 1 N- Terminal Propeptide (P1NP) at Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Description: P1NP, a marker of bone formation was assayed from plasma. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
micrograms per liter (mcg/L)
  Study Baseline: number analyzed (Participants) | 30
  Study Baseline | 44.3960 (15.7898)
  Change at Week 26: number analyzed (Participants) | 30
  Change at Week 26 | -0.6947 (9.8577)
  Change at Week 52: number analyzed (Participants) | 29
  Change at Week 52 | 2.0917 (12.4906)
  Change at Week 78: number analyzed (Participants) | 27
  Change at Week 78 | 3.6133 (16.5480)
  Change at Week 104: number analyzed (Participants) | 28
  Change at Week 104 | 1.6300 (12.2829)
  Change at Week 130: number analyzed (Participants) | 28
  Change at Week 130 | 0.1675 (14.7345)
  Change at Week 156: number analyzed (Participants) | 28
  Change at Week 156 | -1.9043 (11.5887)
  Change at Week 182: number analyzed (Participants) | 28
  Change at Week 182 | 1.6632 (12.1623)
  Change at Week 208: number analyzed (Participants) | 26
  Change at Week 208 | 0.1354 (14.6972)
  Change at Week 234: number analyzed (Participants) | 12
  Change at Week 234 | 3.4467 (12.1002)

23. Primary Outcome: Change From Eliglustat Baseline in Bone Biomarker Level: Procollagen 1 N- Terminal Propeptide (P1NP) at Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Description: P1NP, a marker of bone formation was assayed from plasma. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234 of the current study
Population: Here, "0" signifies that data for this outcome measure (bone biomarker P1NP) was not collected and assessed in Phase 2 and Phase 3 studies, hence the biomarker level was not reported at specified timepoints.
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Change From Current Study Baseline in Bone Biomarker Level: Type 1 Collagen C-Telopeptides (CTx) at Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Description: CTx, a marker of bone resorption was assayed from plasma. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
mcg/L
  Study Baseline: number analyzed (Participants) | 30
  Study Baseline | 0.4540 (0.1827)
  Change at Week 26: number analyzed (Participants) | 30
  Change at Week 26 | -0.0363 (0.1515)
  Change at Week 52: number analyzed (Participants) | 29
  Change at Week 52 | -0.0034 (0.1309)
  Change at Week 78: number analyzed (Participants) | 27
  Change at Week 78 | -0.0041 (0.1696)
  Change at Week 104: number analyzed (Participants) | 28
  Change at Week 104 | 0.0000 (0.1660)
  Change at Week 130: number analyzed (Participants) | 27
  Change at Week 130 | -0.0426 (0.1420)
  Change at Week 156: number analyzed (Participants) | 26
  Change at Week 156 | -0.0738 (0.1294)
  Change at Week 182: number analyzed (Participants) | 28
  Change at Week 182 | 0.0011 (0.2439)
  Change at Week 208: number analyzed (Participants) | 25
  Change at Week 208 | -0.0176 (0.1812)
  Change at Week 234: number analyzed (Participants) | 12
  Change at Week 234 | 0.1200 (0.2150)

25. Primary Outcome: Change From Eliglustat Baseline in Bone Biomarker Level: Type 1 Collagen C-Telopeptides (CTx) at Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234
Description: CTx, a marker of bone resorption was assayed from plasma. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 26, 52, 78, 104, 130, 156,182, 208 and 234 of the current study
Population: Here, "0" signifies that data for this outcome measure (bone biomarker CTx) was not collected and assessed in Phase 2 and Phase 3 studies, hence the biomarker level was not reported at specified timepoints.
Groups:
- Eliglustat: Participants From ENCORE: Participants who completed study GZGD02607 (ENCORE) were included in this current (EFC13781) study. Participants who were CYP2D6 IM, EM and URM received eliglustat 84 mg twice daily and participants who were CYP2D6 PM received eliglustat 84 mg once daily, for duration of minimum 2 years (unless early discontinuation occurred), or until commercial eliglustat was available to participants through reimbursement (up to maximum of 4 years).
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Change From Current Study Baseline in Gaucher Disease Type 1 (GD1) Biomarker Levels: Chitotriosidase at Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: Chitotriosidase biomarker was assayed from plasma. Chitotriosidase biomarker levels for participants who were CYP2D6 non-Ultra Rapid Metabolizers (non-URM) was reported in this outcome measure. For this outcome measure, baseline refers to the study baseline, which was defined as status at study entry.
Time Frame: Study Baseline, Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Population: Analysis was performed on FAS population. Here, "overall number of participants analyzed" = participants evaluable for this outcome measure and "number analyzed" = participants with available data for each specified category. Baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | Eliglustat
Number analyzed (Participants) | 30
nmol/hr/mL
  Study Baseline | 4039.3333 (4441.8462)
  Change at Week 26 | -411.2333 (2486.4359)
  Change at Week 52: number analyzed (Participants) | 29
  Change at Week 52 | -308.6897 (2843.4606)
  Change at Week 78: number analyzed (Participants) | 28
  Change at Week 78 | -492.4286 (3850.9447)
  Change at Week 104: number analyzed (Participants) | 28
  Change at Week 104 | -709.2143 (3274.5604)
  Change at Week 130: number analyzed (Participants) | 28
  Change at Week 130 | -712.4643 (3366.5521)
  Change at Week 156: number analyzed (Participants) | 28
  Change at Week 156 | -367.9286 (3615.7654)
  Change at Week 182: number analyzed (Participants) | 28
  Change at Week 182 | -582.1429 (3386.1815)
  Change at Week 208: number analyzed (Participants) | 26
  Change at Week 208 | -334.1538 (3523.8660)
  Change at Week 234: number analyzed (Participants) | 13
  Change at Week 234 | 411.7692 (1880.7128)

27. Secondary Outcome: Change From Eliglustat Baseline in Gaucher Disease Type 1 (GD1) Biomarker Levels: Chitotriosidase at Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: Chitotriosidase biomarker was assayed from plasma. Chitotriosidase biomarker levels for participants who were CYP2D6 non-URM was reported in this outcome measure. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Time Frame: Eliglustat Baseline, Week 26, 52, 78, 104, 130, 156, 182, 208 and 234 of the current study
Population: Analysis was performed on FAS population. Here, "overall number of participants analyzed" = participants evaluable for this outcome measure and "number analyzed" = participants with available data for each specified category and "0" in number analyzed field signifies that none of the participants had evaluable data at specified timepoint.
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 3
nmol/hr/mL
  Eliglustat Baseline: number analyzed (Participants) | 27 | 2
  Eliglustat Baseline | 9507.9630 (7618.0282) | 2844.5000 (338.7041)
  Change at Week 26: number analyzed (Participants) | 27 | 2
  Change at Week 26 | -6054.5185 (6817.9692) | -122.5000 (2112.1280)
  Change at Week 52: number analyzed (Participants) | 26 | 2
  Change at Week 52 | -6207.9615 (7178.4162) | -405.5000 (2581.6469)
  Change at Week 78: number analyzed (Participants) | 25 | 2
  Change at Week 78 | -6475.0800 (8035.2136) | -1233.0000 (2054.8523)
  Change at Week 104: number analyzed (Participants) | 25 | 2
  Change at Week 104 | -6704.6000 (7658.9433) | -1249.0000 (2186.3742)
  Change at Week 130: number analyzed (Participants) | 25 | 2
  Change at Week 130 | -6663.5200 (7578.2222) | -981.5000 (2724.4824)
  Change at Week 156: number analyzed (Participants) | 25 | 2
  Change at Week 156 | -6335.6000 (7785.3273) | -1181.0000 (2494.6727)
  Change at Week 182: number analyzed (Participants) | 25 | 2
  Change at Week 182 | -6543.0000 (7349.2169) | -933.0000 (2851.0545)
  Change at Week 208: number analyzed (Participants) | 23 | 2
  Change at Week 208 | -6380.3913 (7729.7877) | -1160.5000 (2560.4337)
  Change at Week 234: number analyzed (Participants) | 13 | 0
  Change at Week 234 | -7212.0769 (7757.2285) |

28. Secondary Outcome: Change From Current Study Baseline in GD1 Biomarker Levels: Glucosylceramide (GL-1) at Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: Glucosylceramide (GL-1) biomarker was assayed from plasma. GL-1 biomarker levels for participants who were CYP2D6 non-URM was reported in this outcome measure. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Eliglustat
Number analyzed (Participants) | 30
micrograms per milliliter (mcg/mL)
  Study Baseline | 5.3243 (3.5830)
  Change at Week 26 | -1.7770 (3.8871)
  Change at Week 52: number analyzed (Participants) | 29
  Change at Week 52 | -1.7002 (4.6162)
  Change at Week 78: number analyzed (Participants) | 28
  Change at Week 78 | -1.4000 (4.1376)
  Change at Week 104: number analyzed (Participants) | 28
  Change at Week 104 | -2.0657 (3.5678)
  Change at Week 130: number analyzed (Participants) | 28
  Change at Week 130 | -1.7405 (3.5448)
  Change at Week 156: number analyzed (Participants) | 28
  Change at Week 156 | -1.6073 (3.3841)
  Change at Week 182: number analyzed (Participants) | 28
  Change at Week 182 | -1.7304 (3.8140)
  Change at Week 208: number analyzed (Participants) | 26
  Change at Week 208 | -2.0408 (3.7987)
  Change at Week 234: number analyzed (Participants) | 13
  Change at Week 234 | 0.7691 (2.2570)

29. Secondary Outcome: Change From Eliglustat Baseline in GD1 Biomarker Levels: Glucosylceramide (GL-1) at Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: Glucosylceramide (GL-1) biomarker was assayed from plasma. GL-1 biomarker levels for participants who were CYP2D6 non-URM was reported in this outcome measure. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Time Frame: Eliglustat Baseline, Week 26, 52, 78, 104, 130, 156, 182, 208 and 234 of the current study
Population: Analysis was performed on FAS population. Here, "overall number of participants analyzed" = participants evaluable for this outcome measure and "number analyzed" = participants with available data for each specified category and "0" signifies that none of the participants had evaluable data at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 3
mcg/mL
  Eliglustat Baseline: number analyzed (Participants) | 23 | 3
  Eliglustat Baseline | 11.8304 (3.5804) | 5.9667 (0.9713)
  Change at Week 26: number analyzed (Participants) | 23 | 3
  Change at Week 26 | -8.2095 (3.6233) | -2.2470 (3.7756)
  Change at Week 52: number analyzed (Participants) | 22 | 3
  Change at Week 52 | -8.0970 (4.0568) | -2.9880 (3.3407)
  Change at Week 78: number analyzed (Participants) | 21 | 3
  Change at Week 78 | -7.7498 (3.7788) | -3.1150 (3.5522)
  Change at Week 104: number analyzed (Participants) | 21 | 3
  Change at Week 104 | -8.6111 (3.7016) | -3.6920 (2.8225)
  Change at Week 130: number analyzed (Participants) | 21 | 3
  Change at Week 130 | -8.5354 (3.8700) | -3.2767 (1.8706)
  Change at Week 156: number analyzed (Participants) | 21 | 3
  Change at Week 156 | -8.1772 (3.4306) | -1.8643 (5.6710)
  Change at Week 182: number analyzed (Participants) | 21 | 3
  Change at Week 182 | -8.0321 (3.6982) | -3.9720 (2.0463)
  Change at Week 208: number analyzed (Participants) | 19 | 3
  Change at Week 208 | -8.5976 (3.4497) | -4.2390 (2.2343)
  Change at Week 234: number analyzed (Participants) | 13 | 0
  Change at Week 234 | -7.9463 (3.6203) |

30. Secondary Outcome: Change From Current Study Baseline in GD1 Biomarker Levels: Lyso Glucosylceramide (Lyso-GL-1) at Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: Lyso-GL-1 biomarker was assayed from plasma. Lyso-GL-1 biomarker levels for participants who were CYP2D6 non-URM was reported in this outcome measure. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Eliglustat
Number analyzed (Participants) | 30
nanograms per milliliter (ng/mL)
  Study Baseline: number analyzed (Participants) | 21
  Study Baseline | 114.2429 (89.5197)
  Change at Week 26: number analyzed (Participants) | 21
  Change at Week 26 | -43.8238 (63.2152)
  Change at Week 52: number analyzed (Participants) | 20
  Change at Week 52 | -40.7500 (61.0894)
  Change at Week 78: number analyzed (Participants) | 19
  Change at Week 78 | -30.6711 (71.1072)
  Change at Week 104: number analyzed (Participants) | 19
  Change at Week 104 | -35.5721 (47.2414)
  Change at Week 130: number analyzed (Participants) | 19
  Change at Week 130 | -33.6195 (74.1656)
  Change at Week 156: number analyzed (Participants) | 19
  Change at Week 156 | -27.6795 (72.4469)
  Change at Week 182: number analyzed (Participants) | 19
  Change at Week 182 | -32.3611 (71.9446)
  Change at Week 208: number analyzed (Participants) | 17
  Change at Week 208 | -31.2882 (64.0608)
  Change at Week 234: number analyzed (Participants) | 6
  Change at Week 234 | -45.5100 (31.0448)

31. Secondary Outcome: Change From Eliglustat Baseline in GD1 Biomarker Levels: Lyso Glucosylceramide (Lyso-GL-1) at Week 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: Lyso-GL-1 biomarker was assayed from plasma. Lyso-GL-1 biomarker levels for participants who were CYP2D6 non-URM was reported in this outcome measure. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Time Frame: Eliglustat Baseline, Week 26, 52, 78, 104, 130, 156, 182, 208 and 234 of the current study
Population: Analysis was performed on FAS population. Here, "overall number of participants analyzed" = participants evaluable for this outcome measure and "number analyzed" = participants with available data for each specified category. Here, "0" in overall number analyzed field signifies that biomarker lyso-GL-1 was not assessed in Phase 3 studies, hence the biomarker levels at specified timepoint were not reported for any of the participants who were from previous Phase 3 studies.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 0
ng/mL
  Eliglustat Baseline: number analyzed (Participants) | 9 | 0
  Eliglustat Baseline | 612.2222 (256.6835) |
  Change at Week 26: number analyzed (Participants) | 9 | 0
  Change at Week 26 | -548.3111 (236.1365) |
  Change at Week 52: number analyzed (Participants) | 9 | 0
  Change at Week 52 | -537.1222 (250.8135) |
  Change at Week 78: number analyzed (Participants) | 9 | 0
  Change at Week 78 | -522.6833 (248.3267) |
  Change at Week 104: number analyzed (Participants) | 9 | 0
  Change at Week 104 | -516.3022 (236.9183) |
  Change at Week 130: number analyzed (Participants) | 9 | 0
  Change at Week 130 | -516.9889 (238.9292) |
  Change at Week 156: number analyzed (Participants) | 9 | 0
  Change at Week 156 | -511.6000 (241.2484) |
  Change at Week 182: number analyzed (Participants) | 9 | 0
  Change at Week 182 | -516.5111 (244.4099) |
  Change at Week 208: number analyzed (Participants) | 8 | 0
  Change at Week 208 | -495.3500 (261.1088) |
  Change at Week 234: number analyzed (Participants) | 6 | 0
  Change at Week 234 | -590.8100 (220.5445) |

32. Secondary Outcome: Change From Current Study Baseline in Short Form-36 Health Survey (SF-36) Scores at Weeks 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: The 36-Item Short-Form Health Survey (SF-36) is standardized survey evaluating 8 aspects of functional health and well-being. Physical Component Summary (PCS) with 4 sub-scales: physical function, role limitations due to physical problems, bodily pain, and general health perception; and Mental Component Summary (MCS) with 4 sub-scales: vitality, social function, role limitations due to emotional problems, and mental health. Summations of item scores of the same sub-scale give the sub-scale scores, which are transformed into a range from 0 to 100; 0= worst and 100=best outcome. Both PCS and MCS range from 0 to 100 with higher scores indicating better physical and mental health. For this outcome measure, baseline refers to the current study baseline, which was defined as status at this study (EFC13781) entry.
Time Frame: Study Baseline, Weeks 26, 52, 78, 104, 130, 156, 182, 208 and 234
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
score on a scale
  Study Baseline: PCS | 52.8795 (6.5046)
  PCS: Week 26 | 53.3052 (6.1692)
  PCS: Change at Week 26 | 0.4258 (3.3324)
  PCS: Week 52 | 52.8240 (6.0361)
  PCS: Change at Week 52 | -0.0554 (3.8484)
  PCS: Week 78: number analyzed (Participants) | 29
  PCS: Week 78 | 53.0769 (5.7370)
  PCS: Change at Week 78: number analyzed (Participants) | 29
  PCS: Change at Week 78 | -0.5431 (3.9927)
  PCS: Week 104: number analyzed (Participants) | 29
  PCS: Week 104 | 53.1225 (5.5751)
  PCS: Change at Week 104: number analyzed (Participants) | 29
  PCS: Change at Week 104 | -0.4975 (3.0048)
  PCS: Week 130: number analyzed (Participants) | 29
  PCS: Week 130 | 52.2996 (6.6942)
  PCS: Change at Week 130: number analyzed (Participants) | 29
  PCS: Change at Week 130 | -1.3203 (4.4392)
  PCS: Week 156: number analyzed (Participants) | 29
  PCS: Week 156 | 51.6359 (6.5758)
  PCS: Change at Week 156: number analyzed (Participants) | 29
  PCS: Change at Week 156 | -1.9841 (3.5507)
  PCS: Week 182: number analyzed (Participants) | 29
  PCS: Week 182 | 52.4094 (6.4415)
  PCS: Change at Week 182: number analyzed (Participants) | 29
  PCS: Change at Week 182 | -1.2105 (4.0492)
  PCS: Week 208: number analyzed (Participants) | 29
  PCS: Week 208 | 52.2733 (7.2695)
  PCS: Change at Week 208: number analyzed (Participants) | 29
  PCS: Change at Week 208 | -1.3466 (4.6688)
  PCS: Week 234: number analyzed (Participants) | 13
  PCS: Week 234 | 52.5847 (5.5468)
  PCS: Change at Week 234: number analyzed (Participants) | 13
  PCS: Change at Week 234 | -1.0284 (4.5981)
  Study Baseline: MCS | 49.6223 (11.2360)
  MCS: Week 26 | 51.7497 (9.4775)
  MCS: Change at Week 26 | 2.1274 (5.8293)
  MCS: Week 52 | 50.1502 (11.2198)
  MCS: Change at Week 52 | 0.5279 (8.9388)
  MCS: Week 78: number analyzed (Participants) | 29
  MCS: Week 78 | 51.0151 (10.1117)
  MCS: Change at Week 78: number analyzed (Participants) | 29
  MCS: Change at Week 78 | -0.2412 (5.9877)
  MCS: Week 104: number analyzed (Participants) | 29
  MCS: Week 104 | 50.0147 (12.7162)
  MCS: Change at Week 104: number analyzed (Participants) | 29
  MCS: Change at Week 104 | -1.2415 (7.1779)
  MCS: Week 130: number analyzed (Participants) | 29
  MCS: Week 130 | 51.6144 (10.6866)
  MCS: Change at Week 130: number analyzed (Participants) | 29
  MCS: Change at Week 130 | 0.3582 (5.7170)
  MCS: Week 156: number analyzed (Participants) | 29
  MCS: Week 156 | 51.5030 (10.6347)
  MCS: Change at Week 156: number analyzed (Participants) | 29
  MCS: Change at Week 156 | 0.2468 (7.0860)
  MCS: Week 182: number analyzed (Participants) | 29
  MCS: Week 182 | 52.1595 (9.6141)
  MCS: Change at Week 182: number analyzed (Participants) | 29
  MCS: Change at Week 182 | 0.9033 (6.0446)
  MCS: Week 208: number analyzed (Participants) | 29
  MCS: Week 208 | 49.2308 (11.8064)
  MCS: Change at Week 208: number analyzed (Participants) | 29
  MCS: Change at Week 208 | -2.0254 (7.6197)
  MCS: Week 234: number analyzed (Participants) | 13
  MCS: Week 234 | 47.7470 (12.5183)
  MCS: Change at Week 234: number analyzed (Participants) | 13
  MCS: Change at Week 234 | -3.9989 (8.9392)

33. Secondary Outcome: Change From Eliglustat Baseline in SF-36 Scores at Weeks 26, 52, 78, 104, 130, 156, 182, 208 and 234
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being. PCS with 4 sub-scales: physical function, role limitations due to physical problems, pain, and general health perception; and MCS with 4 sub-scales: vitality, social function, role limitations due to emotional problems, and mental health. Summations of item scores of same sub-scale give the sub-scale scores, which are transformed into range from 0 to 100; 0= worst, and 100=best outcome. Both PCS and MCS range from 0 to 100, higher scores indicating better physical and mental health. For this outcome measure, baseline refers to the eliglustat baseline, which was defined as participant's status at the time of first dose of eliglustat in the previous Phase 2 or Phase 3 study.
Time Frame: Eliglustat Baseline, Weeks 26, 52, 78, 104, 130, 156, 182, 208 and 234 of the current study
Population: Analysis was performed on full analysis population. Here, "number analyzed" = participants with available data for each specified category "0" signifies that none of the participants had evaluable data at the specified timepoint. Data for this outcome measure was planned to be collected and analyzed in reference to eliglustat baseline separately for participants from Phase 2, ENGAGE and EDGE studies (GD treatment naïve participants) and from ENCORE study (participants switched from ERT).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eliglustat: Participants From Phase 2, ENGAGE and EDGE | Eliglustat: Participants From ENCORE
Number analyzed (Participants) | 27 | 4
score on a scale
  Study Baseline: PCS: number analyzed (Participants) | 23 | 4
  Study Baseline: PCS | 43.0578 (6.0372) | 42.7817 (1.4815)
  PCS: Week 26 | 53.0454 (6.0420) | 55.0589 (7.7136)
  PCS: Change at Week 26: number analyzed (Participants) | 23 | 4
  PCS: Change at Week 26 | 9.4479 (9.3442) | 12.2772 (8.2025)
  PCS: Week 52 | 52.8961 (5.8443) | 52.3379 (8.2436)
  PCS: Change at Week 52: number analyzed (Participants) | 23 | 4
  PCS: Change at Week 52 | 9.0581 (8.8189) | 9.5562 (8.8310)
  PCS: Week 78: number analyzed (Participants) | 25 | 4
  PCS: Week 78 | 53.1474 (5.2925) | 52.6363 (9.1001)
  PCS: Change at Week 78: number analyzed (Participants) | 21 | 4
  PCS: Change at Week 78 | 9.6365 (9.2094) | 9.8546 (9.6980)
  PCS: Week 104: number analyzed (Participants) | 25 | 4
  PCS: Week 104 | 52.8224 (5.5216) | 54.9983 (6.3833)
  PCS: Change at Week 104: number analyzed (Participants) | 21 | 4
  PCS: Change at Week 104 | 9.0939 (8.6935) | 12.2166 (7.0338)
  PCS: Week 130: number analyzed (Participants) | 25 | 4
  PCS: Week 130 | 52.2561 (6.0816) | 52.5714 (11.0568)
  PCS: Change at Week 130: number analyzed (Participants) | 21 | 4
  PCS: Change at Week 130 | 8.9364 (9.5735) | 9.7897 (11.8746)
  PCS: Week 156: number analyzed (Participants) | 25 | 4
  PCS: Week 156 | 51.6309 (6.1757) | 51.6671 (9.9228)
  PCS: Change at Week 156: number analyzed (Participants) | 21 | 4
  PCS: Change at Week 156 | 8.1580 (9.4576) | 8.8854 (10.5054)
  PCS: Week 182: number analyzed (Participants) | 25 | 4
  PCS: Week 182 | 52.5222 (5.6686) | 51.7047 (11.3772)
  PCS: Change at Week 182: number analyzed (Participants) | 21 | 4
  PCS: Change at Week 182 | 9.5587 (9.0071) | 8.9229 (12.1080)
  PCS: Week 208: number analyzed (Participants) | 25 | 4
  PCS: Week 208 | 52.4226 (5.9064) | 51.3400 (14.5875)
  PCS: Change at Week 208: number analyzed (Participants) | 21 | 4
  PCS: Change at Week 208 | 9.2886 (9.1756) | 8.5582 (15.2331)
  PCS: Week 234: number analyzed (Participants) | 13 | 0
  PCS: Week 234 | 52.5847 (5.5468) |
  PCS: Change at Week 234: number analyzed (Participants) | 13 | 0
  PCS: Change at Week 234 | 8.7252 (7.2170) |
  Study Baseline: MCS: number analyzed (Participants) | 23 | 4
  Study Baseline: MCS | 41.8312 (8.5951) | 42.4960 (7.0731)
  MCS: Week 26 | 52.7415 (7.3261) | 45.0552 (19.0913)
  MCS: Change at Week 26: number analyzed (Participants) | 23 | 4
  MCS: Change at Week 26 | 9.9441 (8.2305) | 2.5592 (14.2291)
  MCS: Week 52 | 50.5915 (10.9200) | 47.1715 (14.5528)
  MCS: Change at Week 52: number analyzed (Participants) | 23 | 4
  MCS: Change at Week 52 | 8.0060 (8.7063) | 4.6756 (9.2744)
  MCS: Week 78: number analyzed (Participants) | 25 | 4
  MCS: Week 78 | 51.1656 (10.1361) | 50.0740 (11.4453)
  MCS: Change at Week 78: number analyzed (Participants) | 21 | 4
  MCS: Change at Week 78 | 6.2543 (7.5038) | 7.5780 (7.7376)
  MCS: Week 104: number analyzed (Participants) | 25 | 4
  MCS: Week 104 | 51.4510 (10.2052) | 41.0384 (23.4822)
  MCS: Change at Week 104: number analyzed (Participants) | 21 | 4
  MCS: Change at Week 104 | 6.9764 (6.7131) | -1.4576 (18.5758)
  MCS: Week 130: number analyzed (Participants) | 25 | 4
  MCS: Week 130 | 52.5954 (9.4948) | 45.4826 (16.9277)
  MCS: Change at Week 130: number analyzed (Participants) | 21 | 4
  MCS: Change at Week 130 | 7.7807 (6.0885) | 2.9866 (13.2768)
  MCS: Week 156: number analyzed (Participants) | 25 | 4
  MCS: Week 156 | 52.1408 (9.3668) | 47.5165 (18.1409)
  MCS: Change at Week 156: number analyzed (Participants) | 21 | 4
  MCS: Change at Week 156 | 8.0714 (5.6904) | 5.0205 (13.3734)
  MCS: Week 182: number analyzed (Participants) | 25 | 4
  MCS: Week 182 | 52.8180 (8.8447) | 48.0439 (14.5143)
  MCS: Change at Week 182: number analyzed (Participants) | 21 | 4
  MCS: Change at Week 182 | 8.5582 (7.2613) | 5.5479 (9.6766)
  MCS: Week 208: number analyzed (Participants) | 25 | 4
  MCS: Week 208 | 50.0376 (10.3762) | 44.1884 (20.0085)
  MCS: Change at Week 208: number analyzed (Participants) | 21 | 4
  MCS: Change at Week 208 | 5.9449 (7.3056) | 1.6924 (14.9871)
  MCS: Week 234: number analyzed (Participants) | 13 | 0
  MCS: Week 234 | 47.7470 (12.5183) |
  MCS: Change at Week 234: number analyzed (Participants) | 13 | 0
  MCS: Change at Week 234 | 4.0884 (7.5215) |

34. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. A serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the treatment-emergent period (time from the first administration of the investigational medicinal product (IMP) to the last administration of the IMP + 5 days).
Time Frame: From the first administration of the IMP to the last administration of the IMP + 5 days (up to 4 years, or until commercial eliglustat was available to participants through reimbursement or through the compassionate use [expanded access] program)
Population: Analysis was performed on FAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 31
Participants
  TEAEs | 19
  TESAEs | 4

ADVERSE EVENTS:
Time Frame: Time from the first administration of the IMP to the last administration of the IMP + 5 days (up to 4 years, or until commercial eliglustat was available to participants through reimbursement or through the compassionate use [expanded access] program)
Description: Reported adverse events (AEs) are TEAEs i.e. AEs that developed, worsened, or became serious during the treatment-emergent period (time from the first administration of the IMP to the last administration of the IMP + 5 days). Analysis was performed on FAS population.
Arm/Group | Eliglustat
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 4/31
Other Adverse Events (participants affected / at risk) | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eliglustat (N=31)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eliglustat (N=31)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (3)
Human Chorionic Gonadotropin Increased (Investigations) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (3)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT02536755/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT02536755/SAP_001.pdf